CLINICAL TRIAL: NCT01945164
Title: Single Patient Treatment Study for the Use of XL999 Administered Intravenously to a Subject With Advanced Malignancies Previously Enrolled in Study XL999-900
Brief Title: XL999 Administered Intravenously to a Subject With Advanced Malignancies
Status: No longer available | Type: Expanded Access
Sponsor: John Sarantopoulos (Other)
Responsible Party: Sponsor-Investigator, John Sarantopoulos, Principal Investigator, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Other Study IDs: CTRC 10-08; HSC20100312H (Other: UTHSCSA IRB)
Record Dates: First submitted 2012-12-07; First posted 2013-09-18 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Advanced Malignancy
Keywords: XL999; Advanced Malignancy

INTERVENTIONS:
Drug: XL999 — The treatment will consist of 4-week cycles in which the subject will receive XL999 administered as a 4-hour IV infusion every other week. The subject will continue to receive 4-week cycles of XL999 in the absence of progressive disease, unacceptable drug-related toxicity, and as long as the drug is available.

SUMMARY:
Cancer is a worldwide clinical and economic problem. Conventional approaches to treating cancer include surgery, radiotherapy, and cytotoxic chemotherapy as single modalities or as combined therapies. Recently, targeted therapies including antibodies and small molecule inhibitors have also demonstrated clinical benefit. It is now possible to study different genetic lesions involved in cancer types due to advances in genomic methodologies. The investigational drug in this study, XL999 inhibits multiple receptor tyrosine kinases, including VEGF receptor (VEGFR2/KDR), platelet derived growth factor receptors (PDGFRβ), fms-like tyrosine kinase receptor 3 (FLT3), fibroblast growth factor receptors (FGFR1, FGFR3), RET, and KIT, and thus, interferes with multiple cellular processes simultaneously and will likely have effects on the integrity of tumor neovasculature and angiogenesis. Together with the ability to induce a novel cell cycle arrest, the spectrum of activities that XL999 exhibits may reduce both tumor cell proliferation and angiogenesis in the clinic.

The rationale and purpose of this maintenance study is to allow a subject receiving clinical benefit from XL999 to continue treatment.

ELIGIBILITY:
Inclusion Criteria:

* The subject is eligible to continue to receive XL999 in the absence of progressive disease and unacceptable XL999-related toxicity.

Exclusion Criteria:

* Progressive disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2010-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Sarantopoulos, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Cancer Therapy and Research Center at UTHSCSA, San Antonio, Texas, United States